CLINICAL TRIAL: NCT04409041
Title: Oral Low-Dose Naltrexone in the Treatment of Lichen Planopilaris and Frontal Fibrosing Alopecia; an Uncontrolled Open-label Prospective Study
Brief Title: Oral Low-Dose Naltrexone for Lichen Planopilaris and Frontal Fibrosing Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201908021
Record Dates: First submitted 2020-05-22; First posted 2020-06-01 (Actual); Results first posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-11

CONDITIONS: Lichen Planopilaris; Frontal Fibrosing Alopecia
MeSH Terms: conditions — Lichen Planus | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-dose naltrexone group (Experimental): All participants were prescribed low-dose naltrexone at 3mg oral daily.
  Interventions: Drug: Low-Dose Naltrexone

INTERVENTIONS:
Drug: Low-Dose Naltrexone — Based on the promising evidence, we propose using low-dose naltrexone at a daily dose of 3mg to treat lichen planopilaris and frontal fibrosing alopecia. The patients would be continued on their other medications for these conditions. The study would be open-label, so all participants would receive the low-dose naltrexone. Patients would be seen at 0,3,6 and 12 months to monitor their progress.

SUMMARY:
Oral naltrexone was initially FDA approved to treat opioid use disorder and alcohol dependence at doses from 50-100mg/day. At lower doses of 1-5mg/day, naltrexone has been used off-label with success in treatment of several dermatologic conditions including the scarring hair loss disease lichen planopilaris. A recent case series of four patients with lichen planopilaris and a subtype, frontal fibrosing alopecia, treated with oral low-dose naltrexone at 3mg daily showed reduction of itch, clinical evidence of inflammation of the scalp, and of disease progression. There were no reported adverse events.

Based on the promising evidence, we propose using low-dose naltrexone at a daily dose of 3mg to treat lichen planopilaris and frontal fibrosing alopecia. The patients would be continued on their other medications for these conditions. The study would be open-label, so all participants would receive the low-dose naltrexone. Patients would be seen at 0,3,6 and 12 months to monitor their progress.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or greater
* clinically or histologically confirmed diagnosis of lichen planopilaris or frontal fibrosing alopecia

Exclusion Criteria:

* known allergy or hypersensitivity to naltrexone
* patients with concurrent use of opioids
* active depression, schizophrenia, and bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group (Low-dose Naltrexone): Everyone enrolled received low-dose naltrexone at 3mg oral daily.
Period: Overall Study
Arm/Group | Treatment Group (Low-dose Naltrexone)
Started | 43
Completed | 26
Not Completed | 17

BASELINE CHARACTERISTICS:
Population: 43 patients enrolled.
Arm/Group | Treatment Group (Low-dose Naltrexone)
Number analyzed (Participants) | 43
Age, Continuous [Median (Standard Deviation); unit: years] | 65 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-Reported Itch
Description: 0-10 scale for itch. Lower scores are better outcome. A change between two time points is reported at 12 months.
Time Frame: 12 months
Population: Per protocol group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group (Low-dose Naltrexone)
Number analyzed (Participants) | 26
units on a scale | -0.33 [-1.08 to 0.41]

2. Primary Outcome: Change in Investigator Rated Erythema
Description: 0-3 scale for erythema. Higher scores are worse. A change between two time points is reported at 12 months.
Time Frame: 12 months
Population: Per protocol group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group (Low-dose Naltrexone)
Number analyzed (Participants) | 26
units on a scale | -0.93 [-1.32 to -0.53]

3. Primary Outcome: Patient Reported Burning/Pain
Description: Patient reported burning/pain on 0-10 scale. Higher values are worse. A change between two time points is reported at 12 months.
Time Frame: 12 months
Population: Per protocol group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low-dose Naltrexone Group
Number analyzed (Participants) | 26
units on a scale | -0.50 [-1.02 to 0.02]

4. Primary Outcome: Change in Investigator Rated Scale
Description: Investigator assessed outcome of scale on 0-3 scale. Higher numbers are worse. A change between two time points is reported at 12 months.
Time Frame: 12 months
Population: Per protocol group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low-dose Naltrexone Group
Number analyzed (Participants) | 26
units on a scale | -0.33 [-0.72 to 0.07]

ADVERSE EVENTS:
Time Frame: 12 months.
Description: Adverse events collected for the 12-month study period. There was no control group. 34 patients received at least one dose of naltrexone and were assessed for adverse events (however only 26 patients had follow up assessments that allowed them to be included in the efficacy analysis for primary outcomes).
Arm/Group | Treatment Group (Low-dose Naltrexone)
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 2/34
Other Adverse Events (participants affected / at risk) | 10/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (Low-dose Naltrexone) (N=34)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (Low-dose Naltrexone) (N=34)
vivid dreams (Nervous system disorders) | 7 (7)
headache (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT04409041/Prot_SAP_000.pdf